CLINICAL TRIAL: NCT02840539
Title: A Phase 2 Trial to Evaluate the Efficacy of Bortezomib, Cytarabine, and Dexamethasone in Patients With Relapsed or Refractory Mantle Cell Lymphoma
Brief Title: Trial of Bortezomib, Cytarabine, and Dexamethasone in Mantle Cell Lymphoma
Acronym: BATMAN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Consortium for Improving Survival of Lymphoma (Other)
Responsible Party: Principal Investigator, YOUNGIL KOH, Associate Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUH-1602-153-747
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Mantle Cell Lymphoma
Keywords: Mantle cell lymphoma; Bortezomib; Cytarabine
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Bortezomib; Cytarabine; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Bortezomib, Cytarabine, Dexamethasone, Pegteograstim
  Interventions: Drug: Bortezomib, Cytarabine, Dexamethasone, Pegteograstim

INTERVENTIONS:
Drug: Bortezomib, Cytarabine, Dexamethasone, Pegteograstim — Bortezomib: 1.3mg/m2 per day, SC (mixed with normal saline 1.4ml) on day 1, 4, 8, and 11 of each 28-day cycle
  Cytarabine: 1.5g/m2 per day, IV (in the vein) over 3 hours on day 2 and 3 of each 28-day cycle for subjects aged less than 65 and 1g/m2 with the same route and schedule for those aged 65 or older
  Dexamethasone: 20mg per day, IV (in the vein) or PO on day 1, 4, 8, and 11 of each 28-day cycle
  Pegfilgrastim: 6mg once, SC on day 13 of each 28-day cycle Number of cycles: 6 unless progression or unacceptable toxicity develops within 6 cycles
  Other Names: Protezomib, Cytarabine, Dexamethasone, Neulapeg

SUMMARY:
The purpose of this study is to determine whether bortezomib, cytarabine, and dexamethasone are effective in the treatment of relapsed or refractory mantle cell lymphoma after 1 to 3 lines of previous treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed mantle cell lymphoma
* Relapse or progression after 1-3 lines of previous chemotherapy with or without immunologic agents
* ECOG performance status 2 or less
* Adequate hematologic, hepatic, and renal function i. White blood cells ≥ 3,000 /ul ii. Absolute neutrophil count ≥ 1,000 /ul iii. Platelets ≥ 50,000 /ul iv. Hemoglobin ≥ 9.0 g/dL v. Total bilirubin < 2 times upper limit of normal vi. AST, ALT < 2.5 times upper limit of normal vii. Serum creatinine < 1.5 times upper limit of normal

Exclusion Criteria:

* Previously treated with 4 or more lines of chemotherapy with or without immunologic agents
* Previously treated with bortezomib
* Treated with a cytarabine-containing regimen as the last line and within 6 months before registration
* Other cancer diagnosed within 5 years before registration
* Uncontrolled symptomatic CNS involvement of mantle cell lymphoma
* Uncontrolled systemic infection
* Inherited immunodeficiency disease or AIDS
* Pregnancy
* Breast-feeding
* Peripheral neuropathy of grade 3 or higher
* Other health conditions considered to be inappropriate for this trial in the primary physician's opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Overall response | within 28 days after the last cycle of treatment
  Lugano classification

SECONDARY OUTCOMES:
Complete response | within 28 days after the last cycle of treatment
  Lugano classification
Overall survival | 5 years
  Interval from registration to death from any cause
Progression-free survival | 5 years
  Interval from registration to progression or death from any cause

OTHER OUTCOMES:
Quality of life | within 28 days after the last cycle of treatment
  EORTC QLQ-C30
Toxicity | within 28 days after the last cycle of treatment
  NCI CTCAE version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Youngil Koh, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Demographics, baseline characteristics, response, survival data

REFERENCES:
- [Background] Robak T, Huang H, Jin J, Zhu J, Liu T, Samoilova O, Pylypenko H, Verhoef G, Siritanaratkul N, Osmanov E, Alexeeva J, Pereira J, Drach J, Mayer J, Hong X, Okamoto R, Pei L, Rooney B, van de Velde H, Cavalli F; LYM-3002 Investigators. Bortezomib-based therapy for newly diagnosed mantle-cell lymphoma. N Engl J Med. 2015 Mar 5;372(10):944-53. doi: 10.1056/NEJMoa1412096. PMID 25738670
- [Derived] Shin J, Lee JY, Lee GW, Kim WS, Park Y, Do YR, Kim DS, Kim KH, Choi YS, Byun JM, Hong J, Kim I, Yoon SS, Koh Y. Phase II study of bortezomib, cytarabine and dexamethasone in relapsed or refractory mantle cell lymphoma. Br J Haematol. 2023 Sep;202(6):e54-e57. doi: 10.1111/bjh.18965. Epub 2023 Jul 5. No abstract available. PMID 37408333